CLINICAL TRIAL: NCT03749681
Title: Neuroendocrine Tumors of Patients Aged of 75 y or Over in the West of France
Brief Title: Neuroendocrine Tumors of Old Patients in the West of France
Acronym: TANGO
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: University Hospital, Brest (Other)
Collaborators: Novartis (Industry)
Responsible Party: Sponsor
Other Study IDs: TANGO (29BRC18.0013)
Record Dates: First submitted 2018-04-05; First posted 2018-11-21 (Actual); Last update posted 2018-11-21 (Actual); Status verified 2018-03

CONDITIONS: Neuroendocrine Tumors
Keywords: Neuroendocrine Tumors; 75 y and over patients; Oncogeriatric follow-up; Oncologic care
MeSH Terms: conditions — Neuroendocrine Tumors

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Neuroendocrine cancer remains a poorly known entity. Comprehensive treatment is multidisciplinary involving surgery, radiological and nuclear medicine, and medical. A national network for the management of sporadic and hereditary malignant neuro-ENdocrine Tumor (RENATEN) is in charged of coordinating this specific care. This is part of the French National Cancer INstitute (INCa) Rare Cancer Plan.

The project is in the form of an analysis of elderly population (75 years or over) with a diagnosis of neuroendocrine cancer in the western part of the France (Brittany, Pays de Loire, Normandy, Center and a part of New Aquitaine areas) representing a population of more than 12 millions of inhabitants. Oncogeriatric evaluations, specialized meetings, ...would be analysed in order to improve the care of rare cancer patients.

ELIGIBILITY:
Inclusion Criteria:

* 75 years old or over at the time of diagnosis
* Patient with G1/G2/G3 neuroendocrine tumor diagnosed by pathological analysis
* Patient whose medical file was examined by RENATEN (National Network for the treatment of neuro-ENdocrine sporadic and hereditary disease Tumor) meetings or other multidisciplinary consultation meeting between 01/01/2014 and 31/12/2017
* Patient with care in private and public centers in the West of France

Exclusion Criteria:

* Patient with cancer other than a neuroendocrine tumor
* Patient with a G4 neuroendocrine tumor
* Patient who has objected to the study and collection of his medical data
* Refusal of participation

Min Age: 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Study Population: Elderly patients with a neuroendocrine tumor whose medical file was analysed by RENATEN group between 2014 and 2017 in 4 western regions
Sampling Method: Non-Probability Sample
Enrollment: 306 (Estimated)
Dates: Start 2018-12 (Estimated); Primary Completion 2020-03-28 (Estimated); Study Completion 2020-03-28 (Estimated)

PRIMARY OUTCOMES:
Tumor description : localization of the tumor (digestive or others) provided by scan or anatomopathologic report | 03/31/2020
  statistical analysis (%)
All anticancer treatment description in neuroendocrine tumors of 3 specific histological grade (G1, 2 or 3) | 03/31/2020
  statistical analysis (%)
Histology, differentiation status | 03/31/2020
  qualitative description (text)
mitotic index and proliferation idex of the tumor | 03/31/2020
  statistical analysis (%)
Response rate | 03/31/2020
  statistical analysis (%)
progression free survival | 03/31/2020
  statistical analysis (months) with Kaplan meier analysis; data provided by the medical file
overall survival | 03/31/2020
  statistical analysis (months) with Kaplan meier analysis; data provided by the medical file

CONTACTS AND LOCATIONS:
Locations (1):
- CHRU de Brest, Brest, France

IPD SHARING:
Plan to Share IPD: No